CLINICAL TRIAL: NCT03612362
Title: Effect of Improved "Injera" Baking Stove Intervention on Household Air Pollution and Childhood Acute Respiratory Infection Prevention: A Cluster Randomized Controlled Trial In Northwest Ethiopia
Brief Title: Impact of Improved "Injera" Baking Stove Use on Childhood Acute Respiratory Infection Prevention in Northwest Ethiopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bahir Dar University (Other)
Responsible Party: Principal Investigator, Mesafint Molla, Assistant Professor at School of Public Health, College of Medicine and Health Sciences, Bahir Dar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 088/18-04; U1111-1215-1090 (Registry Identifier: Universal Trial Number)
Record Dates: First submitted 2018-07-24; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Acute Respiratory Infection; Pneumonia Childhood
Keywords: Acute Respiratory Infection, Household Air Pollution

STUDY DESIGN:
Intervention Model Description: Cluster randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Improved "Injera" Baking Biomass Stove (Experimental): 2750 eligible households with in 50 randomly selected clusters/"Gotes" are allocated into the improved "Injera" backing stove intervention arm.
  Interventions: Device: Improved "Injera" Baking Biomass Stove
- Control arm (No Intervention): Similarly 2750 eligible households with in 50 randomly selected clusters/Gotes will continue to use the traditional "Injera" baking biomass stove and will be used as control arm.

INTERVENTIONS:
Device: Improved "Injera" Baking Biomass Stove — Replacing of the Ethiopian traditional "Injera" baking biomass stove with improved baking biomass stove, the well-known commercially distributed type of baking stove in Ethiopia, will be the intervention for this study. Control HHs will continue to use the traditional baking biomass stove. Concerning intervention duration, since the life span of the Ethiopian improved baking stove is about 5 years, the length of the intervention period will be one year to account for seasonal factors that have major effect on both ARI incidence & HAP level in Ethiopia as well as to maintain a balance between achieving a sufficiently long follow-up period for outcome measurements & suitably short follow-up period to decrease attrition.
  Arms: Improved "Injera" Baking Biomass Stove

SUMMARY:
In Ethiopia, great majorities (95%) of households rely on solid biomass fuels such as wood, muck, crop residues, and charcoal burned in highly polluting stoves to meet the basic household energy needs with its severe health consequences due to emission of toxic indoor air pollutants. Correspondingly, household air pollution (HAP) from biomass fuel use is now estimated to be responsible for nearly 3.5 million premature deaths annually, with the highest disease burdens experienced by countries in sub-Saharan Africa. HAP ranks as the highest environmental risk factors to premature deaths globally and 2nd leading risk factor next to childhood underweight in most of sub-Saharan Africa countries as well as 3rd leading risk factor of disease next to childhood underweight, and suboptimal breastfeeding in Ethiopia.

Usually prevention efforts aimed at reducing HAP and related health burdens have been focused on the use of energy efficient cookstoves. There is, however, rigorous lack of evidence in Ethiopia or in other similar settings whether it is possible to achieve adequate HAP reduction and improve health with locally made energy efficient baking stoves from a public health point of view. Particularly, the popular Ethiopian energy efficient "Injera" baking stove has not been researched through stove trial inquiry. Therefore, research studies are required in Ethiopia on health benefits achieved when households adopt energy efficient baking stoves. In view of that, cluster randomized controlled trial will be employed with experimental study design for one year to test the effectiveness of the Ethiopian improved "Injera" baking stove intervention on reducing HAP and childhood acute respiratory infection (ARI) through comparing equal size groups of children before and after part of households received an improved "Injera" baking stove.

Accordingly, the proposed stove trial aims to address an important research gap by determining whether the Ethiopian improved "Injera" baking biomass stove intervention can adequately reduce HAP exposure to prevent childhood acute respiratory infection. With this objective, the proposed stove trial will test the hypothesis that there is a statistically significant difference in HAP levels and incidence of childhood ARI when using traditional versus improved "Injera" baking stove in Northwest Ethiopia

DETAILED DESCRIPTION:
1. Study area:

   The implementation of the study project has been started among rural and urban communities of Mecha Health & Demographic Surveillance System (MHDSS) Site in Northwest Ethiopia. MHDSS site is a field research center established by Bahir Dar University (BDU) to conduct field researches & support major graduate level research projects principally. The field research center is located at 525 km far away from the capital city of Ethiopia, Addis Ababa, towards Northwest. This field research center has been selected as study area in light of the following particular rationales:
   * Relevance of the project to the community in terms of current biomass fuel use, climatic diversity & local acceptability of the improved stove intervention
   * Strategic research importance of the locality to achieve the mission's of BDU to be one of the ten premiere research universities in Africa by the year 2025.
   * Opportunities to be benefited from the existing field research infrastructures of MHDSS
   * Availability of local collaborators with experience of improved stove technology transfer
   * Availability of improved baking stove initiatives already operating in the study area
   * Good field experience of investigators at the study area
2. Study design:

   Cluster randomized controlled study will be employed to test the effectiveness of improved "Injera" baking biomass stove intervention in reducing both household air pollution (HAP) & childhood acute respiratory infection (ARI) incidences through comparing children living in households (HHs) with different baking stoves over one year follow-up period. With this study design, HAP & childhood ARI outcomes will be measured before the improved baking stove is installed and again after part of the HHs received an improved baking stove. The overall study procedures will involve the following three major phases:
   * Base line data collection using HH interview and air monitoring methods.
   * Installing improved "Injera" baking biomass stove in the main cooking area of the intervention HHs to be used as primary baking stove at least for one year.
   * Consecutive data collection using the HH interview method every 2 weeks and measure the new amounts of indoor particulate matter in the main cooking area using standard HAP monitoring device every 3 months for one year.
3. Sample size:

   For the primary outcome, the sample size was calculated by applying the two-sample comparison of proportions formula using STATA with equal participants in both arms considering 21% proportion of childhood ARI, detectable difference of 20%, & two-tailed alpha of 0.05, power of 80%, intra-cluster correlation coefficient (Ƿ) value of 0.01, coefficient of variation of 0.6 for cluster sizes, 55 average number of children within each cluster (m') and over sampling of 10%; the required sample size with cluster randomization becomes about 2750 within 50 clusters per arm. Similarly, for the secondary outcome, the sample size was calculated by considering detectable difference of 60% in mean indoor PM2.5 concentration (µg/m3), correlation coefficient (Ƿ) of 0.5 for indoor PM2.5 measurement variations in biomass using HHs, 2-sided alpha of 0.05, power of 80% and 55 average number of children within each cluster (m'), 0.6 coefficient of variation for cluster sizes and over sampling of 10%; the required sample size becomes about 990 within 18 clusters per arm. Thus, among the HHs included in the primary outcome study, only part of the HHs will be included for the secondary outcome study.
4. Sampling method:

   Using cluster sampling technique, clusters/"Gotes" will be selected randomly to represent the total population & then all HHs with under 4 years old child with in the selected clusters will be included. A cluster is defined as the small village, termed as "Gote" for rural or "Ketena" for urban settings in Amharic (both national & local language), used as the smallest unit of enumeration area by Ethiopian national census. According to the update data report of MHDSS at the end of 2017, each cluster/"Gote" includes about 55 average number of children. To set the randomisation list in advance based on eligibility criteria, the sampling frame (list of HHs with children less than 4 years old) is established form the MHDSS update report data. Finally, the selected HHs will be identified for data collection using the specific MHDSS house number & the youngest child equal or less than 4 years old will be recruited for study from each HH. In situations where there are 2 or more under-four children living in the same HH, only the youngest child will be included in the study.
5. Participant recruitment:

   To facilitate the participant enrolment process, community sensitization will be conducted through public communications during local gatherings & regular health development army (HDA) meetings as well as through home visit by health & agricultural extension workers to let people know that childhood ARI & HAP studies will be carried out. The actual participants will be recruited at HH level by field health workers during baseline survey after ensuring whether the HHs meet the eligibility criteria. When HH meets the eligibility criteria, the study will be explained to parent/s of the index child & they will be asked whether the HH is willing to participate in the studies or not. When both parents agreed to be involved, the field staff will administer a written consent form in local language.
6. Participant allocation:

   An independent epidemiologist was performed the allocation to control & intervention arms which will be revealed after all baseline measurements have been completed as well as all study HHs recruited & assigned to their respective arm to ensure allocation concealment.
7. Intervention adherence and compliance monitoring strategies:

   To avoid the potential detrimental effects of non-adherence, a variety of strategies will be used. In view of that, timely response to trial-related difficulties such as rapid maintenance or replacing of defective stoves will be used as strategy to improve adherence to the intervention protocol. Regarding trial protocol compliance monitoring, visual inspection through unannounced visit of HHs will be conducted to enhance validity of data.
8. Data collection methods:

   For the primary objective, data collection will be carried out by local nurses through face-to-face interview with index child mothers/caregivers using questionnaire & through direct verification whenever essential & possible. After baseline HH survey, the follow up survey will be carried out for one year through HH visits every 2 weeks. Concerning the duration, since seasonal factors typically have a major effect on HAP level in Ethiopia the duration of the follow-up period will be one year to cover the major Ethiopian periods of annual weather changes. Data collection manual containing a detailed description of the questions & other administrative issues will be used to facilitate data collection process. For the secondary objective, baseline HAP exposure (indoor PM2.5 concentration) will be measured in the main cooking area using standard HAP monitoring device and Standard Operating Procedures (SOPs) by trained household air monitoring team. In addition, independent variables data will be collected at baseline through face-to-face interview with index child mothers/caregivers using structured questionnaire. After baseline survey & implementation of improved stove intervention, subsequent indoor PM2.5 concentration measurements & other covariates data collection will be carried out every 3 months for one year.
9. Data handling and analysis:

   All original participant files will be stored in a secured manner for a period of at least 2 years after completion of the study. Data integrity will be enforced through a variety of mechanisms such as double data entry; valid values checks & consistency checks against data already stored in the database (i.e., longitudinal checks). Considering the underlying design of the study, assumptions regarding the inter-relationship between the independent & outcome variables under investigation as well as the repeated & dependent nature of the data, Generalized Estimating Equation modeling method of data analysis will be applied to determine the effect of improved baking stove intervention on both HAP & childhood ARI incidence.
10. Ethical consideration and trial registration:

    The proposal had been reviewed & approved on May 08/2018 by Institutional Ethical Review Board of Bahir BDU. Written informed consent will be obtained from all participants. The informed consent process emphasizes that participation in the study is voluntary & consent to participation can be withdrawn at any time, without giving a reason as well as without affecting their current or future benefits to which the participants are entitled. Moreover, to maintain justice control HHs will be offered improved baking biomass stove at the end of their participation. Whenever ARI illness is occurred, field health workers will refer the child to the nearest health institution for proper treatment.
11. Close-out procedures:

The trial will be terminated at the planned target of one year after the last participant has been randomized or at an earlier or later date if the circumstances necessitate. Regardless of the timing & circumstances of the end of the study, close-out will proceed in 2 stages: the first stage covers the interim period for analysis & documentation of study results which is expected to take about 3 months. The second stage will comprise debriefing of participants & dissemination of study results.

ELIGIBILITY:
Inclusion Criteria:

* Households with children up to 4 years old to ensure a minimum of one year longitudinal data collection before the child's 5th birthday.
* Households who bake "Injera" exclusively with a traditional baking stove

Exclusion Criteria:

* Households who do not have any enclosed main cooking area (kitchen) structure
* Children who will be born during the course of the study

Max Age: 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5500 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Longitudinal proportion of childhood acute respiratory infection as measured by childhood pneumonia status using World Health Organization's Integrated Management of Neonatal and Childhood Illness algorism. | Change from baseline childhood ARI due to Improved "Injera" Baking Stove Intervention will be assessed at one year.
  Childhood acute respiratory infection/pneumonia status will be assessed using standard case recording form by field workers during household visits where the index child mothers/caregivers are asked about ARI signs & symptoms in the preceding two weeks. Moreover, to overcome some of the limitations of the self-reported health data, physical examination of the ill index child will be conducted by field workers trained in World Health Organization's Integrated Management of Neonatal and Childhood Illness algorism.

SECONDARY OUTCOMES:
Household air pollution as measured by concentration of indoor particulate matter with an aerodynamic diameter of less than 2.5 microns (PM2.5) in µg/m3 | Change from baseline HAP (indoor PM2.5 concentration) due to Improved "Injera" Baking Stove Intervention will be assessed at one year.
  To estimate the household level exposure to pollutant for each household enrolled in this longitudinal study, the concentration of PM2.5 will be measured in the main cooking area following Standard Operating Procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Mesafint M. Adane, MPH,BSc.,, Principal Investigator — School of Public Health, College of Medicine and Health Sciences, Bahir Dar University, Ethiopia; Prof. Getu D. Alene, PhD,, Study Chair — Department of Epidemiology and Biostatics, School of Public Health, College of Medicine and Health Sciences, Bahir Dar University, Ethiopia; Dr. Seid T. Mereta, PhD,, Study Director — Department of Environmental Health Science & Technology, School of Public Health, Jimma University
Locations (1):
- "Mecha" Health and Demographic Surveillance System (MHDSS) Site, Bahir Dar University, Bahir Dar, Amhara Regional State, Ethiopia

REFERENCES:
- [Background] Baumgartner J, Smith KR, Chockalingam A. Reducing CVD Through Improvements in Household Energy: Implications for Policy-Relevant Research. Glob Heart. 2012 Sep;7(3):243-7. doi: 10.1016/j.gheart.2012.06.018. No abstract available. PMID 25691487
- [Background] Berhane K, Kumie A, Samet J. Health Effects of Environmental Exposures, Occupational Hazards and Climate Change in Ethiopia: Synthesis of Situational Analysis, Needs Assessment and the Way Forward. Ethiop J Health Dev. 2016;30(1 Spec Iss):50-56. PMID 28867920
- [Background] Bonjour S, Adair-Rohani H, Wolf J, Bruce NG, Mehta S, Pruss-Ustun A, Lahiff M, Rehfuess EA, Mishra V, Smith KR. Solid fuel use for household cooking: country and regional estimates for 1980-2010. Environ Health Perspect. 2013 Jul;121(7):784-90. doi: 10.1289/ehp.1205987. Epub 2013 May 3. PMID 23674502
- [Background] Budds J, Biran, A. & Rouse, J. What's Cooking: a review of the health impacts of indoor air pollution and technical interventions for its reduction. 2001
- [Background] Campbell MK, Fayers PM, Grimshaw JM. Determinants of the intracluster correlation coefficient in cluster randomized trials: the case of implementation research. Clin Trials. 2005;2(2):99-107. doi: 10.1191/1740774505cn071oa. PMID 16279131
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Desalegn B, Suleiman H, Asfaw A. Household fuel use and acute respiratory infections among younger children: an exposure assessment in Shebedino Wereda, Southern Ethiopia. African Journal of Health Sciences. 2011;18(1-2):31-6
- [Background] Edwards R, Hubbard A, Khalakdina A, Pennise D, Smith KR. Design considerations for field studies of changes in indoor air pollution due to improved stoves. Energy for Sustainable Development June 2007;11(2)
- [Background] Energy Sector Mapping and Database Development. Ethiopian Ministry of Water and Energy, 2013a
- [Background] Hemming K, Girling AJ, Sitch AJ, Marsh J, Lilford RJ. Sample size calculations for cluster randomised controlled trials with a fixed number of clusters. BMC Med Res Methodol. 2011 Jun 30;11:102. doi: 10.1186/1471-2288-11-102. PMID 21718530
- [Background] Household cookstove, environment, health, and climate change: a new look at an old problem, The World Bank, The Environment Department (Climate Change). 2011
- [Background] Kernan WN, Viscoli CM, Makuch RW, Brass LM, Horwitz RI. Stratified randomization for clinical trials. J Clin Epidemiol. 1999 Jan;52(1):19-26. doi: 10.1016/s0895-4356(98)00138-3. PMID 9973070
- [Background] Kumie A, Emmelin A, Wahlberg S, Berhane Y, Ali A, Mekonen E, Worku A, Brandstrom D. Sources of variation for indoor nitrogen dioxide in rural residences of Ethiopia. Environ Health. 2009 Nov 18;8:51. doi: 10.1186/1476-069X-8-51. PMID 19922645
- [Background] Kumie A, Samet J, Berhane K. Air Pollution, Occupational Health and Safety, and Climate Change: Findings, research needs and policy implications establishing a GEOHealth Hub for East Africa. Situational analysis and needs assessment for Ethiopia. August 2014
- [Background] Lim SS, Vos T, Flaxman AD, Danaei G, Shibuya K, Adair-Rohani H, Amann M, Anderson HR, Andrews KG, Aryee M, Atkinson C, Bacchus LJ, Bahalim AN, Balakrishnan K, Balmes J, Barker-Collo S, Baxter A, Bell ML, Blore JD, Blyth F, Bonner C, Borges G, Bourne R, Boussinesq M, Brauer M, Brooks P, Bruce NG, Brunekreef B, Bryan-Hancock C, Bucello C, Buchbinder R, Bull F, Burnett RT, Byers TE, Calabria B, Carapetis J, Carnahan E, Chafe Z, Charlson F, Chen H, Chen JS, Cheng AT, Child JC, Cohen A, Colson KE, Cowie BC, Darby S, Darling S, Davis A, Degenhardt L, Dentener F, Des Jarlais DC, Devries K, Dherani M, Ding EL, Dorsey ER, Driscoll T, Edmond K, Ali SE, Engell RE, Erwin PJ, Fahimi S, Falder G, Farzadfar F, Ferrari A, Finucane MM, Flaxman S, Fowkes FG, Freedman G, Freeman MK, Gakidou E, Ghosh S, Giovannucci E, Gmel G, Graham K, Grainger R, Grant B, Gunnell D, Gutierrez HR, Hall W, Hoek HW, Hogan A, Hosgood HD 3rd, Hoy D, Hu H, Hubbell BJ, Hutchings SJ, Ibeanusi SE, Jacklyn GL, Jasrasaria R, Jonas JB, Kan H, Kanis JA, Kassebaum N, Kawakami N, Khang YH, Khatibzadeh S, Khoo JP, Kok C, Laden F, Lalloo R, Lan Q, Lathlean T, Leasher JL, Leigh J, Li Y, Lin JK, Lipshultz SE, London S, Lozano R, Lu Y, Mak J, Malekzadeh R, Mallinger L, Marcenes W, March L, Marks R, Martin R, McGale P, McGrath J, Mehta S, Mensah GA, Merriman TR, Micha R, Michaud C, Mishra V, Mohd Hanafiah K, Mokdad AA, Morawska L, Mozaffarian D, Murphy T, Naghavi M, Neal B, Nelson PK, Nolla JM, Norman R, Olives C, Omer SB, Orchard J, Osborne R, Ostro B, Page A, Pandey KD, Parry CD, Passmore E, Patra J, Pearce N, Pelizzari PM, Petzold M, Phillips MR, Pope D, Pope CA 3rd, Powles J, Rao M, Razavi H, Rehfuess EA, Rehm JT, Ritz B, Rivara FP, Roberts T, Robinson C, Rodriguez-Portales JA, Romieu I, Room R, Rosenfeld LC, Roy A, Rushton L, Salomon JA, Sampson U, Sanchez-Riera L, Sanman E, Sapkota A, Seedat S, Shi P, Shield K, Shivakoti R, Singh GM, Sleet DA, Smith E, Smith KR, Stapelberg NJ, Steenland K, Stockl H, Stovner LJ, Straif K, Straney L, Thurston GD, Tran JH, Van Dingenen R, van Donkelaar A, Veerman JL, Vijayakumar L, Weintraub R, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams W, Wilson N, Woolf AD, Yip P, Zielinski JM, Lopez AD, Murray CJ, Ezzati M, AlMazroa MA, Memish ZA. A comparative risk assessment of burden of disease and injury attributable to 67 risk factors and risk factor clusters in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2224-60. doi: 10.1016/S0140-6736(12)61766-8. PMID 23245609
- [Background] Meinert CL. Clinical Trials: Design, Conduct and Analysis. New York: Oxford University Press. 1986
- [Background] Rehfuess E, Bruce N, Smith K. Solid Fuel Use: Health Effect. In: Nriagu JO (ed.) Encyclopedia of Environmental Health, v 5, pp. 150161 Burlington: Elsevier, 2011. Environmental Health. 2011;5:150161.
- [Background] Smith KR, Dutta K, Chengappa C, Gusain P, Masera O, Berrueta V, et al. Monitoring and evaluation of improved biomass cookstove programs for indoor air quality and stove performance: conclusions from the Household Energy and Health Project. Energy for Sustainable Development. 2007;11(2):5-18
- [Background] Smith KR, Frumkin H, Balakrishnan K, Butler CD, Chafe ZA, Fairlie I, Kinney P, Kjellstrom T, Mauzerall DL, McKone TE, McMichael AJ, Schneider M. Energy and human health. Annu Rev Public Health. 2013;34:159-88. doi: 10.1146/annurev-publhealth-031912-114404. Epub 2013 Jan 16. PMID 23330697
- [Background] Tefera W, Asfaw A, Gilliland F, Worku A, Wondimagegn M, Kumie A, Samet J, Berhane K. Indoor and Outdoor Air Pollution- related Health Problem in Ethiopia: Review of Related Literature. Ethiop J Health Dev. 2016;30(1):5-16. PMID 28890631
- [Background] Welfare Monitoring Survey. Addis Ababa, Ethiopia: Central Statistical Agency, 2011.
- [Derived] Adane MM, Alene GD, Mereta ST, Wanyonyi KL. Effect of improved cookstove intervention on childhood acute lower respiratory infection in Northwest Ethiopia: a cluster-randomized controlled trial. BMC Pediatr. 2021 Jan 4;21(1):4. doi: 10.1186/s12887-020-02459-1. PMID 33397313
- [Derived] Adane MM, Alene GD, Mereta ST. Biomass-fuelled improved cookstove intervention to prevent household air pollution in Northwest Ethiopia: a cluster randomized controlled trial. Environ Health Prev Med. 2021 Jan 4;26(1):1. doi: 10.1186/s12199-020-00923-z. PMID 33397282